CLINICAL TRIAL: NCT03395600
Title: A Randomized Controlled Comparison of Different Dose Combinations of Bupivacaine and Sufentanil on Epidural Analgesia Onset Time and Adverse Reactions During Labor
Brief Title: Onset of Labour Epidural Analgesia With Different Concentration Bupivacaine and Different Doses of Sufentanyl
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Tingting Wang, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TWang20171226
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Pregnant Women Who Requested Epidural Analgesia in the Early Stage of Labor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.1%bupivacaine+10µg sufentanyl (Active Comparator): Epidural labour analgesia was initiated with 10µg sufentanyl along with 5 ml bupivacaine 0.1% as the test dose. After 3 min, 10 ml of 0.1% bupivacaine epidural was injected
  Interventions: Drug: B1S10
- 0.125%bupivacaine+5µg sufentanyl (Active Comparator): Epidural labour analgesia was initiated with 5µg sufentanyl along with 5 ml bupivacaine 0.125% as the test dose. After 3 min, 10 ml of 0.125% bupivacaine epidural was injected
  Interventions: Drug: B125S5
- 0.1%bupivacaine+5µg sufentanyl (Active Comparator): Epidural labour analgesia was initiated with 5µg sufentanyl along with 5 ml bupivacaine 0.1% as the test dose. After 3 min, 10 ml of 0.1% bupivacaine epidural was injected
  Interventions: Drug: B1S5

INTERVENTIONS:
Drug: B1S5 — Women were then placed supine with left uterine displacement. Epidural labour analgesia was initiated with 5µg sufentanyl along with 5 ml bupivacaine 0.1% as the test dose. After 3 min, 10 ml of 0.1% bupivacaine epidural was injected
  Arms: 0.1%bupivacaine+5µg sufentanyl
Drug: B125S5 — Women were then placed supine with left uterine displacement. Epidural labour analgesia was initiated with 5µg sufentanyl along with 5 ml bupivacaine 0.125% as the test dose. After 3 min, 10 ml of 0.125% bupivacaine epidural was injected
  Arms: 0.125%bupivacaine+5µg sufentanyl
Drug: B1S10 — Women were then placed supine with left uterine displacement. Epidural labour analgesia was initiated with 10µg sufentanyl along with 5 ml bupivacaine 0.1% as the test dose. After 3 min, 10 ml of 0.1% bupivacaine epidural was injected
  Arms: 0.1%bupivacaine+10µg sufentanyl

SUMMARY:
This study aimed to compare the effects of three commonly used combination doses on the onset time and adverse reactions.

DETAILED DESCRIPTION:
Epidural block is widely used as an analgesic method during labor. During epidural anaesthesia, lipophilic opioids such as sufentanil, are often combined with local anesthetics to prolong the duration of analgesia and improve the analgesic effect. However, dose combinations of local anesthetics and opioids, especially in the initial loading dose, vary greatly from hospital to hospital and often depend upon the different routines adopted by anesthesiologists. In clinical practice, there are still some controversy about opioid dose selection in terms of analgesic onset time and adverse reactions.

In this study, three combinations of bupivacaine and sufentanil were chosen, commonly used in the clinic, and extended the observation period to 24 hours after delivery. We hypothesized that increasing the concentration of local anesthetic, rather than increasing the dose of sufentanil, would achieve a faster analgesic effect with minimal adverse effects on the mother and fetus. To test our hypothesis, our primary outcome was to compare the times of analgesia onset of the three combinations, and the secondary outcomes were to compare the effects on maternal and infant adverse reactions.

ELIGIBILITY:
Inclusion Criteria:patients ASA physical status 1 or 2; early labour (cervical dilation 5 cm or less); singleton fetus; gestational age > 36 weeks; and normal fetal heart rate (FHR) tracing. -

Exclusion Criteria:severe preeclampsia;antepartum haemorrhage; ASA 3 or more; chronic pain; substance abuse;contraindications to epidural analgesia; allergies to local anaesthetics or fentanyl; body mass index (BMI) over 40; and previous administration of opioid analgesia within 24 h.

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 56 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
the time to achieve effective analgesia | 30 min
  We defined the onset of analgesia as the time from the start of the injection to the time when the NPRS score was reduced to at least half of the original score.

SECONDARY OUTCOMES:
Sensory block, maternal side effects (pruritus, hypotension, sedation，motor block and decreased fetal heart rate) were recorded at 5-min intervals for 30 min. sedation) | 30min
time from the first PCA bolus, patient satisfaction, type of delivery, fever, establishment of breast feeding and LATCH score within 24 h, cumulative dosage of sufentanil/bupivacaine, time from bolus to delivery. | delivery 24h

CONTACTS AND LOCATIONS:
Overall Officials: Shaoqiang Huang, PhD, Study Chair — Department of Anaesthesia, Obstetrics & Gynecology Hospital, Fudan University
Locations (1):
- Ethics Committee of The Obstetrics and Gynecology Hospital, Fudan University,, Shanghai, China